CLINICAL TRIAL: NCT01878175
Title: Functional Movement Retraining After Hip Arthroplasty in Veterans: Pilot Study
Brief Title: Functional Movement Retraining After Hip Replacement
Acronym: FMR-THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O1033-P
Record Dates: First submitted 2013-06-05; First posted 2013-06-14 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Arthroplasty, Replacement, Hip; Veterans; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional Movement Retraining (Experimental): 15-week rehabilitation / exercise intervention, including visits at the Durham VA medical center, in-home with clinical personnel, and via telephone. The intervention is tailored to participants' post-operative functional status, particularly unilateral balance asymmetries. The exercise program will focus on three areas: lower extremity mobility (ankle, knee and hip), muscle stability (quadriceps and gluteal muscle strength) and functional movement patterns (lower extremity focus). Participants will be instructed to perform their prescribed stretching exercises daily and strengthening exercises three times per week (on non-consecutive days).
  Interventions: Behavioral: Functional Movement Retraining

INTERVENTIONS:
Behavioral: Functional Movement Retraining — 15-week rehabilitation / exercise intervention, including visits at the Durham VA medical center, in-home with clinical personnel, and via telephone. The intervention is tailored to participants' post-operative functional status, particularly unilateral balance asymmetries. The exercise program will focus on three areas: lower extremity mobility (ankle, knee and hip), muscle stability (quadriceps and gluteal muscle strength) and functional movement patterns (lower extremity focus). Participants will be instructed to perform their prescribed stretching exercises daily and strengthening exercises three times per week (on non-consecutive days).

SUMMARY:
Total hip arthroplasty (THA) is a common surgical procedure among Veterans. It is most often used to treat hip osteoarthritis, which is more common among Veterans than the general population. Some patients continue to experience functional limitations after THA, and studies have shown that these patients still tend to put greater loads on the opposite leg, which can increase the risk of developing osteoarthritis in that leg. One likely reason for these post-surgical limitations is that rehabilitation is very minimal following this procedure. This project will involve development and preliminary testing of a functional movement retraining program, designed to help Veterans improve their function and biomechanics after THA. The project will also develop processes for delivering this program in Veterans' homes, to increase accessibility.

DETAILED DESCRIPTION:
Rehabilitation following total hip arthroplasty (THA) is limited in scope, and some patients continue to exhibit functional limitations, as well as loading asymmetries that place them at risk for developing osteoarthritis in contralateral joints. The purpose of this study is to collect preliminary data to support a larger project that will examine the effectiveness of a 12-session functional movement retraining (FMR) program for Veterans following THA. A novel aspect of the FMR program is that it focuses not only on improving overall function but also normalizing side-to-side asymmetries in balance and strength via patient-specific tailoring of exercises. The program also involves telerehabilitation processes to improve access.

Participants will be n=15 patients scheduled for THA at the Durham VAMC, identified from electronic medical records. Participants will complete assessments pre-operatively, then approximately 6-weeks post-THA, at which time FMR program will begin. The 12 FMR sessions will optimally be delivered twice weekly for 6 weeks. However, to account for missed visits, the investigators will allow for 9 total weeks to complete the 12 sessions. Therefore follow-up assessments will be scheduled at 15-weeks post-THA for all participants. FMR sessions will be a combination of: 1.) in-person, on-site visits and telephone contacts with a licensed physical therapist and 2.) in-home telehealth visits by a telehealth technologist or physical therapy assistant. The FMR program will focus on improving lower extremity mobility, muscle stability and functional movement patterns. Participants will be instructed to perform a series of stretching exercises daily and strengthening exercises three times weekly. Exercises for each patient will be tailored according to results of the Lower Quarter Y-Balance Test (conducted at baseline and mid-way through the program), which assesses asymmetries between limbs and between anterior vs. posterior reach. Outcomes will include objective functional measures (timed up-and-go, sit-to-stand, walking speed, stair climb, Lower Quarter Y-Balance Test), self-reported pain and activity limitations (Hip disability and Osteoarthritis Outcome Score), and therapist-assessed function (Harris Hip Score). Basic descriptive statistics will be used to compare changes in each outcome (pre-operative to 15-week post-THA and 6-week post THA to 15-week post-THA) and inform sample size estimates for a larger trial. The investigators will also assess various aspects of program feasibility (recruitment success, adherence, telerehabilitation processes) and collect in-depth qualitative information from both patients and therapists to assess aspects of the intervention that may need to be modified prior to a larger study.

ELIGIBILITY:
Inclusion Criteria:

- Veteran, Scheduled for hip arthroplasty at Durham, NC VA Medical Center

Exclusion Criteria:

- Dementia or other significant cognitive impairment;

* movement or motor neuron disorders (e.g., Parkinson's Disease, post-stroke neurological deficiencies);
* rheumatoid arthritis,
* fibromyalgia,
* or other systemic rheumatic disease;
* hospitalization for a stroke,
* myocardial infarction,
* heart failure,
* or coronary artery revascularization in the past 3 months;
* psychosis or current, uncontrolled substance abuse disorder;
* any other health conditions determined by the study team to be contraindications to performing the exercise program (e.g., mild home exercises);
* transportation or other limitations that would prevent visits to the Durham VAMC for the retraining program.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Functional Movement Retraining: 15-week rehabilitation / exercise intervention, including visits at VA medical center, in-home with clinical personnel, and via telephone. Intervention is tailored to participants' post-operative functional status, particularly unilateral balance asymmetries. The exercise program focuses on lower extremity mobility, muscle stability and functional movement patterns. Participants will be instructed to perform their prescribed stretching exercises daily and strengthening exercises three times per week.
Period: Overall Study
Arm/Group | Functional Movement Retraining
Started | 15
Completed | 13
Not Completed | 2
Not completed — Developed contraindicated health problem | 2

BASELINE CHARACTERISTICS:
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (6.6)
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Hip Disability and Osteoarthritis Outcomes Score (HOOS) - Activities of Daily Living Scale
Description: The HOOS is a validated outcome measure in patients with painful hip conditions. It contains 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and hip related Quality of life (QOL). The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. Change was defined as pre-intervention minus post-intervention. Therefore a negative change score indicates improvement over time.
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Individuals who completed the HOOS ADL scale at 6 weeks and 15 weeks. Two participants were withdrawn from the study before 15 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 13
units on a scale | -6.00 (6.37)

2. Primary Outcome: Change in Hip Disability and Osteoarthritis Outcomes Score (HOOS) - Pain Scale
Description: as for outcome 1
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed the HOOS pain subscale at 6 weeks and 15 weeks. Two participants were withdrawn from the study before 15 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 13
units on a scale | -2.12 (9.78)

3. Primary Outcome: Change in Hip Disability and Osteoarthritis Outcomes (HOOS) Score - Sport Subscale
Description: as for outcome 1
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed the HOOS Sport subscale at 6 weeks and 15 weeks. Two participants were withdrawn from the study before 15 weeks, and one additional participant did not complete all items on this subscale at both time points and therefore could not be given a score, per scale scoring instructions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 12
units on a scale | -20.8 (23.89)

4. Primary Outcome: Change in Hip Disability and Osteoarthritis Outcomes (HOOS) Score - Symptom Subscale
Description: as for outcome 1
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed the HOOS Symptoms subscale at 6 weeks and 15 weeks. Two participants were withdrawn from the study before 15 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 13
units on a scale | -2.69 (10.33)

5. Primary Outcome: Change Hip Disability and Osteoarthritis Outcomes (HOOS) - Quality of Life Subscale
Description: as for outcome 1
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed the HOOS Quality of Life scale at 6 weeks and 15 weeks. Two participants were withdrawn from the study before 15 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 13
units on a scale | -9.13 (22.48)

6. Secondary Outcome: Change in Satisfaction With Physical Function Questionnaire
Description: This is a validated 5-item questionnaire that assesses patients' satisfaction with their ability to complete basic functional tasks that are often affected by lower extremity osteoarthritis (OA), including stair-climbing, walking, doing housework (light and heavy), and lifting and carrying. The scale range is -15 to +15, with higher scores indicating more satisfaction with function. Change was defined as post-intervention minus pre-intervention. Therefore a positive change score indicates improvement over time.
Time Frame: Change between Pre-intervention (post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed the measure at baseline and 15 weeks. Two participants were withdrawn before 15 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 13
units on a scale | 4.14 (1.63)

7. Secondary Outcome: Global Assessment of Hip Symptom Change
Description: We will use the Patient Global Impression of Change scale to evaluate participants' perspectives on overall change in their joint pain in their (one) operative hip during the study period. This single-item measure asks participants to describe their change in pain on a rating scale with the following 13 options: a little worse, somewhat worse, moderately worse, a good deal worse, a great deal worse, a very great deal worse, about the same, a little better, somewhat better, moderately better, a good deal better, a great deal better, a very great deal better. The total scale range is -6 to +6. Negative scores indicate greater perceived improvement.
Time Frame: 15 weeks (post-intervention)
Population: Number of participants who completed this measure at 15 week follow-up. Two participants were withdrawn from the study before 15 weeks, and two additional participants did not complete this item at the 15 week follow up assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 11
units on a scale | -5.09 (0.83)

8. Secondary Outcome: Change in Objective Functional Test: Timed Get Up-and-go
Description: The timed get up-and-go test has demonstrated excellent reliability and correlates well with other standard measures such as gait speed, self-report and clinical report indices of function, and is predictive of who can safely ambulate. This test requires the participants to stand from a standard arm chair, walk 3 meters and then return to sitting in the same chair. Participants are asked to complete this as quickly and safely as possible, without the use of an assistive device. Change was defined as pre-intervention minus post-intervention. Therefore a positive change score indicates improvement over time.
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed this test at both 6 weeks and 15 weeks. Two participants were withdrawn from the study before 15 weeks, and one additional participant did not complete this assessment at both time points.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 12
seconds | 1.23 (5.56)

9. Secondary Outcome: Change in Objective Functional Test: Sit to Stand
Description: The Sit-to-Stand Test has been reported to be a good indicator of postural control, fall risk, lower-extremity strength, and disability. During the sit-to-stand test participants will be asked to place their arms across their chest and keep their feet flat on the floor. They will then be asked to stand up and sit down 5 times as fast as they can. This will be repeated twice and the scores will be averaged for analysis. Change was defined as pre-intervention minus post-intervention. Therefore a positive change score indicates improvement over time.
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed this test at 6 and 15 weeks. Two participants were withdrawn from the study before 15 weeks, and two additional participants did not complete this test at both time points.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 11
seconds | -0.55 (2.33)

10. Secondary Outcome: Change in Objective Functional Test: Walking Speed
Description: Gait speed is a global measure of disability and function and has been correlated with disease processes, fitness level, activities of daily living, and emotional states. In addition, gait speed is an imperative measure for integration to safe and effective community ambulatory status, and has been defined as a reflective measure of function. Walking speed will be determined as the average walking speed over a 3 meter walk. Participants will be asked to walk down a 10 meter walkway 7 times (while wearing standard footwear) to have their walking speed monitored using infrared photocells, while speed is monitored over the middle 3 meters. These seven trials will be averaged in order to determine walking speed at each of the three visits. Change was defined as pre-intervention minus post-intervention. Therefore a negative change score indicates improvement over time.
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed this test at 6 weeks and 15 weeks. Two participants were withdrawn from the study before 15 weeks, and one additional participant did not complete this test at both time points.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 12
m/sec | 0.05 (0.30)

11. Secondary Outcome: Change in Objective Functional Test: Stair Climbing
Description: The task of stair climbing has been found to be sensitive to change with interventions in individuals with knee OA. This measures the time it takes a participant to ascend and descend a flight of 12 steps (each step 18 cm high and 28 cm deep). Participants will be asked to complete the test as quickly as they felt safe and comfortable. The use of one handrail will be allowed if necessary, but patients will be encouraged to minimize their use of the handrail. One practice trial will be performed and the average of two additional tests will be used for analysis. The use of an assistive device will be allowed only if the subject will be unsafe or cannot complete the test without the use of the device. Change was defined as pre-intervention minus post-intervention. Therefore a positive change score indicates improvement over time.
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed this measure at 6 weeks and 15 weeks. Two participants were withdrawn from the study before 15 weeks, and one additional participant did not complete this test at both time points.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 12
seconds | 3.56 (7.65)

12. Secondary Outcome: Change in University of California Los Angeles (UCLA) Activity Questionnaire
Description: The UCLA scale shows a strong correlation with the other measures (r = -0.35 to 0.56 for THA; r = -0.55 to 0.23 for TKA) and discriminates between insufficiently and sufficiently active patients undergoing THA and TKA. The UCLA scale has good reliability, provides high completion rate, and shows no floor effects. It seems to be the most appropriate scale for assessment of physical activity levels in patients undergoing total joint arthroplasty. The UCLA scale is a simple scale ranging from 1 to 10. The patient indicates her or his most appropriate activity level, with 1 defined as 'no physical activity, dependent on others' and 10 defined as 'regular participation in impact sports.' Change was defined as pre-intervention minus post-intervention. Therefore a negative change score indicates improvement over time.
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who completed the test at 6 weeks and 15 weeks. Two participants were withdrawn from the study before 15 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 13
units on a scale | -0.38 (1.80)

13. Secondary Outcome: Change in Harris Hip Score (HHS)
Description: The HHS is the most widely used physician- or therapist-assessed measure of hip function following THA and associated rehabilitation. Although the HHS has also been used in a patient-report format, in this study we will obtain this measure via therapist report, to complement the patient-reported outcomes described above. This measure covers the domains of pain (severity and effects on activities and need for pain medication, function (daily activities and gait), deformity (hip flexion, adduction, internal rotation, and extremity length discrepancy) and range of motion (hip flexion, abduction, internal and external rotation, and adduction). The HHS includes 10 items, with a total score range of 0-100; higher scores indicating better function. The HHS has been shown to be a reliable and valid measure of hip function. Change was defined as pre-intervention minus post-intervention. Therefore a negative change score indicates improvement over time.
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 13
units on a scale | -10.5 (15.67)

14. Secondary Outcome: Change in Lower Quarter Y-balance Test (YBT-LQ)
Description: The YBT-LQ is a test of dynamic balance in unilateral stance . It will be administered to all patients who pass a clearance test, which consists of being able to stand on one leg for 10 seconds. The YBT-LQ is performed for both left and right limbs. Any trial that is failed will be repeated with a maximum of 4 additional trials to be performed in each reach direction, anterior, posterior, and lateral. NOTE: Only although 13 participants began the clearance test at both time points, only 5 participants were able to pass the clearance test required to do the YBT-LQ at 6 weeks. Therefore we have not provided a change score for YBT-LQ since this would involve a very small number of participants, and we are concerned about validity of the results that would be presented since those who completed the test at 6 weeks may be a biased sample. We therefore provide the difference (post minus pre) in the # of participants who completed the clearance test at 15 weeks (9) vs. 6 weeks (5).
Time Frame: Change between Pre-intervention (6 weeks post-surgery) to post-intervention (15 weeks post-surgery)
Population: Number of participants who performed the clearance test for the YBT-LQ at both 6 weeks and 15 weeks.
Measure: Number; unit: Number of participants
Arm/Group | Functional Movement Retraining
Number analyzed (Participants) | 13
Number of participants | 4

ADVERSE EVENTS:
Time Frame: Participants' duration of study participation (approximately 15 weeks following surgery)
Arm/Group | Functional Movement Retraining
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Movement Retraining (N=15)
Inpatient Hospitalization (Psychiatric disorders) | 1 (1) — Not oriented to time and place, possible alcohol withdrawal, anxiety, depression.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Movement Retraining (N=15)
Emergency Room Visit (Injury, poisoning and procedural complications) | 1 (1) — Staple left in hip after replacement, removed
Emergency Room Visit (Infections and infestations) | 1 (1) — Urinary tract infection
Emergency Room Visit (Immune system disorders) | 1 (1) — Food allergy / hives
Emergency Room Visit (Cardiac disorders) | 1 (1) — Hypertension, also blood saturation of surgical wound following surgery
Emergency Room Visit (Musculoskeletal and connective tissue disorders) | 1 (1) — Ankle pain
Emergency Room (Injury, poisoning and procedural complications) | 2 (2) — Fall
Doctor Visit (Injury, poisoning and procedural complications) | 1 (1) — Fall
Emergency Room Visit (General disorders) | 1 (1) — Participant notified study team that he was having swelling in legs and was going to the ER; cancelled study visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes